CLINICAL TRIAL: NCT00130611
Title: B-type Natriuretic Peptide for Acute Shortness of Breath EvaLuation (BASEL) Study - Private Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BASEL III - Private Practice; PP00B-102853/1; 04.001; 287/03
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Dyspnea
Keywords: heart failure; cost effectiveness; BNP; private practice; Acute dyspnoea
MeSH Terms: conditions — Dyspnea; Heart Failure | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BNP blinded therapy (Placebo Comparator): Clinical treatment without knowledge of BNP levels
  Interventions: Other: Clinical examination
- BNP guided therapy (Experimental): Clinical treatment based on clinical examination and BNP-levels
  Interventions: Other: BNP measurement; Other: Clinical examination

INTERVENTIONS:
Other: BNP measurement
  Arms: BNP guided therapy
Other: Clinical examination

SUMMARY:
Cost-effective management of heart failure and pulmonary disease is of paramount importance. Unfortunately, the rapid and accurate differentiation of heart failure from other causes of dyspnea in private practice is challenging. B-type natriuretic peptide (BNP) levels are significantly higher in patients with congestive heart failure as compared to patients with dyspnea due to other causes. As a simple, non-expensive assay easily applicable in private practice is available, rapid measurement of BNP might be very helpful in establishing or excluding the diagnosis of heart failure in patients presenting with acute dyspnea in private practice.

The aim is to test the hypothesis that a BNP guided diagnostic strategy would improve the evaluation and management of patients presenting with acute dyspnea to physicians in private practice and thereby reduce total cost of diagnosis and treatment.

The primary endpoint is total medical cost within 3 months.

DETAILED DESCRIPTION:
Background: Most patients with dyspnea primarily consult physicians in private practice. Heart failure and pulmonary disease are "epidemic" disorders and account for the majority of cases of dyspnea. There are approximately 24 million individuals in the United States with chronic obstructive pulmonary disease and another 10 million persons suffer from asthma. These illnesses generate in excess of 17 million physician office visits a year at a cost of over $10.4 billion. In addition, there are nearly 1.5 million new cases of heart failure in North America and Europe every year. The total direct cost of care for heart failure exceed $38 billion in the United States per year. Therefore, cost-effective management of these diseases is of paramount importance. Unfortunately, the rapid and accurate differentiation of heart failure from other causes of dyspnea in private practice is challenging. The symptoms of heart failure may be nonspecific, and signs are not sensitive enough and considerably overlap with those of pulmonary disease. In addition, signs of volume overload take time to evolve and may be completely absent in patients with acute heart failure.

B-type natriuretic peptide (BNP) is a neurohormone secreted from the cardiac ventricles in response to ventricular volume expansion and pressure overload. BNP levels are significantly higher in patients with congestive heart failure as compared to patients with dyspnea due to other causes. Recently, the researchers were able to show that the use of BNP levels significantly improves the management of patients with acute dyspnea in the emergency department. As a simple, non-expensive assay easily applicable in private practice is available, rapid measurement of BNP might also be very helpful in establishing or excluding the diagnosis of heart failure in patients presenting with acute dyspnea in private practice.

Aim: To test the hypothesis that a BNP guided diagnostic strategy would improve the evaluation and management of patients presenting with acute dyspnea to physicians in private practice and thereby reduce total cost of diagnosis and treatment.

Primary endpoint: Total medical cost within 3 months. Secondary endpoints: Hospitalisation, time interval to the initiation of the most appropriate therapy, 3-month mortality, dyspnea (NYHA) at 3 months, 12-month mortality, 12-month total medical cost, cost-effectiveness.

Patients and Methods: The trial is designed to enrol 250 patients presenting with acute dyspnea to physicians in private practice. Patients will be randomly assigned 1:1 into a control group using evaluation of patients according to local standards without the use of BNP (or other natriuretic peptides) and to a BNP group with early testing for BNP by a rapid point-of-care assay during the first consultation in each private practice.

Expected results: It is the researchers' hypothesis that a BNP guided diagnostic strategy will improve the evaluation and management and thereby reduce total cost of diagnosis and treatment.

Significance: Given the significant morbidity associated with dyspnea, as well as the enormous expenses associated with heart failure and pulmonary disease, BNP testing could represent a major advance in clinical medicine. In addition, BNP testing in the appropriate clinical setting may prove very helpful in the attempts to reduce cost of health care to society without reducing (but possibly increasing) the quality of health care.

ELIGIBILITY:
Inclusion Criteria:

* Acute dyspnoea is the main symptom

Exclusion Criteria:

* Age <18 years
* Obvious traumatic cause
* Severe renal dysfunction (serum creatinine > 250 umol/l)
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-01; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Total medical cost within 3 months | 3 months

SECONDARY OUTCOMES:
Hospitalisation | 1 month
Time interval to the initiation of the most appropriate therapy | 1 month
therapy | 1 month
3-month mortality | 3 month
Dyspnea (New York Heart Association [NYHA]) at 3 months | 3 months
12-month mortality | 12 months
12-month total medical cost | 12 months
Cost-effectiveness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (9):
- Private practices of Baden-Wuertemberg, Freiburg im Breisgau, Freiburg, Germany
- Switzerland (8):
  - Private Practices of Kanton Basel-Landschaft, Basel-Landschaft, Basel-Landschaft
  - Private Practices of Kanton Basel Stadt, Basel, Basel
  - Private practices of Kanton Aargau, Aarau, Canton of Aargau
  - Private Practice of Kanton Schwyz, Altendorf, Canton of Schwyz
  - Private practices of Kanton Solothurn, Solothurn, Canton of Solothurn
  - Private practices of Kanton St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Private Practices of Kanton Graubünden, Chur, Chur
  - Private practices in Kanton Obwalden, Sarnen, Sarnen

REFERENCES:
- [Background] Mueller C, Scholer A, Laule-Kilian K, Martina B, Schindler C, Buser P, Pfisterer M, Perruchoud AP. Use of B-type natriuretic peptide in the evaluation and management of acute dyspnea. N Engl J Med. 2004 Feb 12;350(7):647-54. doi: 10.1056/NEJMoa031681. PMID 14960741
- [Derived] Burri E, Hochholzer K, Arenja N, Martin-Braschler H, Kaestner L, Gekeler H, Hatziisaak T, Buttiker M, Fraulin A, Potocki M, Breidthardt T, Reichlin T, Socrates T, Twerenbold R, Mueller C. B-type natriuretic peptide in the evaluation and management of dyspnoea in primary care. J Intern Med. 2012 Nov;272(5):504-13. doi: 10.1111/j.1365-2796.2012.02552.x. Epub 2012 Jun 12. PMID 22550938
- See also: Related Info — http://www.dyspnea.ch